CLINICAL TRIAL: NCT05999929
Title: Implementation of the Memory Support System: A Feasibility Study
Brief Title: Memory Support System Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bruyère Health Research Institute. (Other)
Collaborators: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: M16-23-024
Record Dates: First submitted 2023-08-03; First posted 2023-08-21 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment
Keywords: Cognition; Intervention; French
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Memory Support System participants (Experimental)
  Interventions: Behavioral: Memory Support System

INTERVENTIONS:
Behavioral: Memory Support System — The MSS is a two-page-per-day, pocket-sized calendar/note-taking system with three sections: (a) events; (b) to do's; and (c) journaling for logging important things to be remembered (e.g., news about family/friends). MSS training consists of ten 1-hour sessions delivered over two or six weeks, starting 7-10 days after baseline assessment.

SUMMARY:
The purpose of this study is to determining the feasibility of providing the Memory Support System (MSS) to individuals with mild cognitive impairment (MCI) and their partners at a clinic in Ontario, Canada. This will involve a) collecting information from patients referred to the a memory clinic and geriatric day hospital about the patient's interest in and the patient's preferred method to administer the MSS; and b) a cost analysis related to implementation of the MSS. The study will also measure efficacy outcomes of the MSS regarding program adherence as well as to self-reported IADLs, self-efficacy for memory, quality of life, mood, anxiety, and caregiver burden among a sample of individuals with MCI and their care partners

DETAILED DESCRIPTION:
A survey will be created and sent out to participants with MCI who have expressed interest in participating in research and have been seen at a memory clinic or geriatric day hospital after the initiation of the study. The survey will consist of a Likert scale and open questions related to patient interest in and preferred length of MSS administration and preference for in-person versus virtual administration.

During and after collection of the survey data, a sample of 20 individuals with MCI (ages ≥50) and their care partners will undergo MSS training.

At enrollment in the MSS training, participants with MCI and their care partners will complete measures of cognitive and functional status. Participants and partners will also complete measures of treatment adherence, IADLs, self-efficacy for memory, quality of life, mood, anxiety, and caregiver burden at baseline, treatment end, and 8-week follow-up. Participants will complete the MSS training consisting of ten 1-hour sessions delivered over two or six weeks, starting 7-10 days after initial assessment. Training will be offered in English or French. After the intervention, participants and their partners will complete a semi-structured interview, seeking suggestions for improving the MSS, teaching curriculum, and intervention logistics.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of single or multi-domain MCI
* Clinical Dementia Rating global (CDR) score of ≤ 0.5
* Montreal Cognitive Assessment score of ≥18
* available contact with a care partner ≥ 2 times weekly
* absence or stable intake of nootropic(s) for ≥ 3 months

Exclusion Criteria:

* visual/hearing impairment and/or history of reading or written inability/disability sufficient to interfere with MSS training
* concurrent participation in another related clinical trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Interest in completion of MSS training | From study start date up to 19 months.
  Percentage of participants that complete the feasibility survey and agree or strongly agree with the statement that they are interested in completing MSS training.

SECONDARY OUTCOMES:
Adherence to French Memory Support System Intervention | One week after starting the treatment (MSS intervention), at completion of the treatment - on average 6 weeks, and at 8 week follow-up after treatment end.
  Change from adherence scores from one week after starting treatment (MSS intervention) at treatment end and at 8 weeks after the treatment end. Using an adherence scale from 0 to 10, with 10 being highest and a cut-off score of ≥ 7 points suggesting adherence with the MSS.
Center for Epidemiologic Studies Depression Scale | Baseline, at completion of the treatment - on average 6 weeks, and at 8 week follow-up after treatment end.
  Change from baseline scale scores at treatment end and at 8 weeks after treatment end. Depression screening scale using Likert scale. Total score of 0-60 points, with higher scores signifying a worse outcome (higher levels of depression).
Everyday Cognition questionnaire. | Baseline, at completion of the treatment - on average 6 weeks, and at 8 week follow-up after treatment end.
  Change from baseline scale scores at treatment end and at 8 weeks after treatment end. Self report measure of performance based instrumental activities of daily living. Total score of 23-92, with higher scores indicating a worse outcome.
Functional Assessment Questionnaire | Baseline, at completion of the treatment - on average 6 weeks, and at 8 week follow-up after treatment end.
  Change from baseline scale scores at treatment end and at 8 weeks after treatment end. Informant based report of performance of instrumental activities of daily living. Total score of 0-30, with higher scores indicating a worse outcome (higher level of dependence).
Quality of Life in Alzheimer Disease | Baseline, at completion of the treatment - on average 6 weeks, and at 8 week follow-up after treatment end.
  Change from baseline scale scores at treatment end and at 8 weeks after treatment end. Self report quality of life scale. Total score of 13-52, with higher scores indicating a better outcome (better quality of life).
State-Trait Anxiety Inventory by the Resources for Enhancing Alzheimer's Caregiver Health project | Baseline, at completion of the treatment - on average 6 weeks, and at 8 week follow-up after treatment end.
  Change from baseline scale scores at treatment end and at 8 weeks after treatment end. Self report anxiety scale. Total score of 10-40 with higher scores indicating a worse outcome (higher level of anxiety).
Chronic Disease Self-efficacy Scale | Baseline, at completion of the treatment - on average 6 weeks, and at 8 week follow-up after treatment end.
  Change from baseline scale scores at treatment end and at 8 weeks after treatment end. Selected questions related to memory and cognition from self report scale. Total score of 9-90 with higher scores indicating a better outcomes (higher feeling of self-efficacy).
Caregiver Burden Inventory Short-Form | Baseline, at completion of the treatment - on average 6 weeks, and at 8 week follow-up after treatment end.
  Change from baseline scale scores at treatment end and at 8 weeks after treatment end. Informant based scale of level of caregiver burden. Total score of 0-48 with higher scores indicating a worse outcome (higher level of burden).

CONTACTS AND LOCATIONS:
Overall Officials: Neil Thomas, MD, Principal Investigator — Bruyère Health Research Institute.; Octavio Santos, PhD, Principal Investigator — Ottawa Hospital Research Institute, Bruyère Health Research Institute
Locations (1):
- Bruyère Health Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from the study may be shared with other researchers within the HABIT consortium. Data that may be shared will include the results of the feasibility survey and the scores from the baseline, treatment end and 8 week follow up outcome measures collected from participants who complete MSS training.
Supporting Information: CSR
Time Frame: Data will be available after the end date of the study and kept indefinitely.
Access Criteria: Upon request that is approved by the study principal investigators.